CLINICAL TRIAL: NCT03627689
Title: Molekule for Allergic Rhinitis/Asthma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accural
Sponsor: Molekule (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Molekule-052018
Record Dates: First submitted 2018-07-02; First posted 2018-08-13 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Asthma; Allergic Rhinitis; Allergic Conjunctivitis
Keywords: asthma; environmental intervention; allergies; air purifier
MeSH Terms: conditions — Asthma; Rhinitis, Allergic; Conjunctivitis, Allergic; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active air purifier arm (Experimental): Active portable air purifier for 1 month at bedside
  Interventions: Other: Active air purifier in respiratory allergies/asthma
- Sham air purifier arm (Sham Comparator): Placebo portable air purifier for 1 month at bedside
  Interventions: Other: Sham air purifier

INTERVENTIONS:
Other: Active air purifier in respiratory allergies/asthma — Continuous use of air purifier to improve allergies and asthma control
  Arms: Active air purifier arm
Other: Sham air purifier — control arm
  Arms: Sham air purifier arm

SUMMARY:
Exposure to airborne allergens and pollutants is linked to symptom severity of allergies, asthma and other respiratory problems. In this study an air purifier using photo-electrochemical oxidation technology (PECO) will be used in the home environment of study participants. The investigator will assess the reduction of symptoms from allergic rhinitis/conjunctivitis and asthma.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of the portable PECO air purifier in reducing symptoms from allergic rhinitis and asthma. Using a randomized, double blinded placebo, controlled trial we will be then able to assess if there are any changes after the use of the PECO air purifier after completing an initial baseline survey & comparing to the exit survey. This is a double-blind study, which means that neither the participant nor the investigator knows which device is being used until after the trial is over.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic allergic rhinitis and/or conjunctivitis by history
2. History of adult asthma requiring medications now or in the past
3. Age ≥18
4. CARAT score less than 24

Exclusion Criteria:

1. Participant is <18 years-old
2. Use of systemic corticosteroids within 14 days of study initiation
3. Treatment with biologic agents or allergen immunotherapy
4. Treatment with other immunomodulators (cyclosporine, azathioprine, hydroxychloroquine, etc)
5. Sensitive to fan sound or blue/purple light at night time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Control of Allergic Rhinitis and Asthma Test (CARAT) score | 4 weeks
  CARAT will measure the change in control scores of respiratory allergies and asthma.
  Scale 0 (Worse control of allergy and asthma) to 30 (Best control of allergy and asthma). The higher score the better control of allergy and asthma.
  There are 10 individual questions, scoring from 0-3.

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil G Rao, MD, Principal Investigator — Molekule
Locations (1):
- Molekule, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT03627689/Prot_000.pdf